CLINICAL TRIAL: NCT05865522
Title: Evaluation of the Effects of Classical Massage to Trapezius Muscle and Foot in Fibromyalgia Patients
Brief Title: Massage of the Trapezius Muscle and Foot in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Erkal (Other)
Responsible Party: Sponsor-Investigator, Emre Erkal, PhD Student, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EmreTez
Record Dates: First submitted 2023-04-25; First posted 2023-05-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Massage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Trapezius Massage Group (Experimental): The patients inTrapezius Group will be given classical massage to the trapezius muscle for 6 weeks, 2 sessions per week (12 sessions in total) by the researcher in the physical therapy unit.
  Patients in trapezius groups will be questioned about their pain with VAS once a week throughout the study. Pain follow-up of the patients in trapezius massage will be performed 48 hours after the massage.
  Interventions: Other: Trapezius Massage
- Foot Massage Group (Experimental): The patients in Foot Group will be given foot massage for 6 weeks, 2 sessions per week (12 sessions in total) by the researcher in the physical therapy unit.
  Patients in foot groups will be questioned about their pain with VAS once a week throughout the study. Pain follow-up of the patients in Foot Massage Group will be performed 48 hours after the massage.
  Interventions: Other: Foot Massage
- Control Group (No Intervention): Patients in Control Group will not receive massage. Patients in control groups will be questioned about their pain with VAS once a week throughout the study.

INTERVENTIONS:
Other: Trapezius Massage — The patients in Trapezius Massage Group will be given classical massage to the trapezius muscle for 6 weeks, 2 sessions per week (12 sessions in total) by the researcher in the physical therapy unit.
  Arms: Trapezius Massage Group
Other: Foot Massage — The patients in Foot Massage Group will be given foot massage for 6 weeks, 2 sessions per week (12 sessions in total) by the researcher in the physical therapy unit.
  Arms: Foot Massage Group

SUMMARY:
Objective: The aim of this study is to evaluate the effect of classical massage on pain, fibromyalgia severity and quality of life in fibromyalgia patients.

Material and Method: The research will be carried out with 75 patients with fibromyalgia who refer to Artvin State Hospital Physical Therapy and Rehabilitation outpatient clinic. The patients will be grouped in 3 through simple randomization: trapezius group , foot group and control group. In the physical therapy unit, the patients in trapezius group will receive a total of 12 sessions of trapezius massage, 2 sessions per week for 6 weeks; the patients in foot group will receive a total of 12 sessions of foot massage, 2 sessions per week for 6 weeks and control group will not receive massage. Patient information form, VAS pain scale, Revised Fibromyalgia Impact Questionnaire and SF 36 Quality of Life Scale will be used to collect data. Chi-square paired t test, Wilcoxon test, one-way analysis of variance and Kruskal Wallis test will be used in the analysis of data.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic disease characterized by widespread musculoskeletal pain associated with a range of somatic symptoms such as fatigue, sleep disturbance, and somatic and cognitive symptoms.

The aim of this study is to evaluate the effect of classical massage on pain, fibromyalgia severity and quality of life in fibromyalgia patients.

The research will be carried out with 75 patients with fibromyalgia who refer to Artvin State Hospital Physical Therapy and Rehabilitation outpatient clinic. The patients will be grouped in 3 through simple randomization: trapezius group, foot group and control group. Fibromyalgia patients coming to the Physical Therapy and Rehabilitation Unit will be met and informed about the research. Written informed consent will be obtained from patients who agree to participate in the study. VAS will be applied to each patient coming to the outpatient clinic and their fulfilment of the inclusion criteria will be determined. Patient information form, FIQR and SF-36 quality of life scale will be applied.

The patients intrapezius group will be given classical massage to the trapezius muscle for 6 weeks, 2 sessions per week (12 sessions in total) by the researcher in the physical therapy unit.

The patients in foot group will be given foot massage for 6 weeks, 2 sessions per week (12 sessions in total) by the researcher in the physical therapy unit.

Patients in control group will not receive massage. Patients in all three groups will be questioned about their pain with VAS once a week throughout the study.

Pain follow-up of the patients in trapezius massage and foot massage groups will be performed 48 hours after the massage.

Pain Scale, Fibromyalgia Impact Questionnaire and SF36 Quality of Life Scale will be administered to the patients in all groups at the end of 6 weeks (post-test). The final test measurements of the participants in trapezius massage and foot massage groups will be made 48 hours after the massage.

Statistical analyses will be performed using the SPSS (IBM SPSS Statistics 23) package program. Shapiro-Wilk or Kolmogorov-Smirnov goodness of fit tests and graphical methods will be used to test whether the distributions of numerical variables conform to the normal distribution. Descriptive statistics such as mean and standard deviation will be given for numerical variables with normal distribution. For numerical variables that do not show normal distribution, descriptive statistics such as median, interquartile distribution range, minimum and maximum will be given. Categorical variables will be presented with frequency and percentage values. Whether there is a difference between categorical variables will be examined by Chi-square (χ2) test. Whether there is a difference in terms of the measurements taken in the three groups and at the two times will be examined by repeated measures two-way ANOVA, if assumptions are met. If the terms interaction are meaningful, we need to examine them separately between groups and within the group. The difference between the groups will be examined with the appropriate ANOVA or Kruskal-Wallis tests. The difference within each group will be examined with the paired-sample t test or Wilcoxon tests, as appropriate. Measurements will be taken for 6 weeks for the VAS score. Whether there is a difference in VAS score within each group will be examined with one-way analysis of variance or Friedman tests, as appropriate.

Statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria

* 18 years and over,
* Diagnosed with fibromyalgia according to ACR 2010 diagnostic criteria
* VAS Pain score of 5 and above,
* No impediment to massage (advanced COPD, asthma, heart or kidney failure, malignant conditions, febrile diseases and pregnancy),
* The areas to be massaged are free of any problems (rash, redness, lesions, temperature increase, swelling, oedema, bone anomalies and localised infections),
* Not using any analgesic medication in the last 24 hours,
* Not receiving physiotherapy in the last 6 months,
* Patients without communication problems were included. Exclusion Criteria
* Receiving physiotherapy,
* Changing pharmacological treatment regimen,
* The one who doesn't come to massage sessions,
* Patients with undesirable effects (bruising and bruising of the skin, etc.) in the massage area were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire | six week
  The scale, which evaluates the effect of fibromyalgia during the last week, consists of 3 sub-dimensions: function (9 items), general effect (2 items) and symptom (10 items) and a total of 21 questions. Scale questions are scored between 0 and 10 points, with 10 indicating the worst possible situation. The total score for the function sub-dimension (between 0 and 90) is divided by 3, the total score for the impact sub-dimension (between 0 and 20) is not divided, and the total score for the symptom sub-dimension (between 0 to 100) is divided by 2 and sub-dimension scores are obtained. The function sub-dimension of the scale ranges between 0 and 30, the impact sub-dimension ranges between 0 and 20, and the symptom sub-dimension ranges between 0 and 50 points. The total scale score is obtained by adding the sub-dimensions, and it is between 0-100; higher scores indicate higher effect of fibromyalgia
Visual Analog Scale (VAS)-Pain | six week
  Visual Analogue Scale (VAS 0-10) is a straight line used to measure the variability of pain, showing the continuity of pain. There is no pain (0) on one end of this line, and most severe pain (10) on the other end. The intensity of pain is marked on this line. The value found by measuring the place marked on the 10 cm long line with a ruler determines the pain.

SECONDARY OUTCOMES:
SF-36 Quality of Life Scale | six week
  The scale, which is widely used to evaluate the quality of life, includes 36 items and 8 dimensions (physical function, social function, pain, energy, emotional role limitation, physical role limitation, mental health and general perception of health). Each dimension score ranges between 0 and 100. Higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Kiyak, PhD, Study Director — Ataturk University
Locations (1):
- Artvin State Hospital Physical Therapy and Rehabilitation outpatient clinic, Artvin, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No